CLINICAL TRIAL: NCT03920553
Title: Evaluation of the Effect on the Application of Hyaluronic Acid Following Laser-assisted Frenectomy
Brief Title: Hyaluronic Acid Application Following Frenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zeynep Turgut Çankaya, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22.12.2018 18.5/9
Record Dates: First submitted 2019-04-13; First posted 2019-04-19 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-04

CONDITIONS: Frenulum; Hypertrophy, Lip
MeSH Terms: conditions — Hypertrophy; Lymphoid Interstitial Pneumonia | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Preoperatively all patients gargled for 1 min with 0.2% chlorhexidine mouthwash. Local anaesthesia was applied to the area where the surgical procedure was to be applied. Then the frenectomy operation was performed with a continuous 970nm wavelength of the diode laser at power setting of 1,5W for approximately 60 seconds from the base to the apex of the frenum, thereby excising it. No bleeding was observed after the frenectomy performed with laser. Then, commercially available Hiyaluronic acid was topically applied to the relevant area to completely cover the surgical field to the test group. Following the frenectomy performed with laser, no application was made to the control group patients.
  Interventions: Biological: Hyaluronic acid
- Control Group (No Intervention): Preoperatively all patients gargled for 1 min with 0.2% chlorhexidine mouthwash. Local anaesthesia was applied to the area where the surgical procedure was to be applied. Then the frenectomy operation was performed with a continuous 970nm wavelength of the diode laser at power setting of 1,5W for approximately 60 seconds from the base to the apex of the frenum, thereby excising it.

INTERVENTIONS:
Biological: Hyaluronic acid — Topical application of hyaluronic acid following Laser assisted frenectomy
  Arms: Test Group

SUMMARY:
This randomized clinical study aimed to compare the outcomes of the laser-assisted frenectomy with and without topical hyaluronic acid application to evaluate the effect of HA on secondary wound healing after frenectomy surgery.

The study included a total of sytemically healthy 40 patients , with high labial frenulum attachment requiring frenectomy. Following laser-assisted frenectomy operation HA gel was applied to the wound surface in the test group, and no application was made to the control group The HA application was made topically to completely cover the surgical area on days 3, 7, and 14 postoperatively. Photographs of the operation area were taken on days 3, 7, and 14. The changes in the area measurements between the digital images according to the healing periods were calculated on a computer. according to Visual Analogue Scale (VAS) was used to evaluate Patient comfort and pain levels.

DETAILED DESCRIPTION:
the aim of this study was to clinically evaluate the effect on secondary wound healing of the topical application of hyaluronic acid to the surgical field after frenectomy operation performed with laser, through evaluation of the amount of reduction of the wound site and postoperative pain levels.The study included a total of 40 patients who had maxillary high labial frenulum attachment and were planned to undergo frenectomy and met the study inclusion criteria. All the patients were informed about oral hygiene control and attention was paid that optimal oral hygiene was maintained throughout the study. Phase I periodontal treatment was applied to patients where necessary. The area measurements of the wound site formed after frenectomy was taken immediately after the frenectomy and on days 3, 7, and 21 postoperatively. HA gel was applied topically after the frenectomy operation to the test group and not to the control group. All the surgical procedures were performed by the same surgeon.

ELIGIBILITY:
Inclusion Criteria:

* No systemic disease,
* the presence of high labial frenulum attachment diagnosed according to Mirko et al., -periodontally healthy or a requirement for periodontal treatment that would only require removing of dental plaque,
* full mouth plaque score <15%,probing pocket depth <3mm in all teeth
* no history of periodontal surgery.

Exclusion Criteria:

* not meet the optimal level of oral hygiene,
* had any condition that could affect wound healing,
* were pregnant or lactating,
* were cigarette smokers or were takiing any medication that might affect the outcome of the study,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
the change in the wound area surface | the area of the wound surface was assessed at baseline and on days 3,7 and 14 days.
  IMAGEJ software was used for the evaluation of the photographs and measurement of the area. The area unit measurements are determined by the operator and for this study, the unit was determined as mm2. To measure the area in the program, the relevant photograph was uploaded to the photograph file and the area to be measured was drawn with the computer mouse. After setting unit calibration, the area measurement was made automatically and the numerical value obtained was recorded in the Excel program.

CONTACTS AND LOCATIONS:
Overall Officials: zeynep Turgut Çankaya, Principal Investigator — Gazi University
Locations (1):
- Zeynep Turgut Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No